CLINICAL TRIAL: NCT01846689
Title: An Open-label Trial of an Erythropoietin Stimulating System to Determine Increased Red Blood Cell Production in Subjects Diagnosed With Anemia of Chronic Disease
Brief Title: An Open-label Trial to Determine Increased Red Blood Cell Production in Subjects With Anemia of Chronic Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Targeted Medical Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E130426
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Anemia of Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ESS (Experimental): Prescription medical food erythropoietin stimulating system
  Interventions: Drug: ESS (medical food/drug)

INTERVENTIONS:
Drug: ESS (medical food/drug) — Prescription medical food erythropoietin stimulating system

SUMMARY:
The objective of this study is to measure the change in blood values after the administration of an amino acid based erythropoietin stimulating system.

ELIGIBILITY:
Inclusion Criteria:

1. M/F patients 18 years old and over, non-pregnant/lactating
2. Hemoglobin < 10 female,<11 male
3. Ferritin > upper limit of normal for lab indicative of chronic anemia
4. Anemia of chronic disease
5. Crt. < 3.0

Exclusion Criteria:

1. Currently taking other amino acid formulations.
2. Pregnant or unwilling to use adequate birth control for the duration of the study.
3. Excessive alcohol or illicit drug use.
4. Unwilling or unable to sign informed consent.
5. Myocardial infarction within the last 6 months.
6. Patients ever having taken or currently taking an erythropoietin medication.
7. Iron deficiency (add criteria).
8. On dialysis.
9. Malignancy other than non-melanoma skin cancer within the last 5 years. If has such malignancy, must have documentation of no recurrence for at least 5 years.
10. Liver cirrhosis (add criteria).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Hemoglogin/Hematocrit | 28 Days

SECONDARY OUTCOMES:
Red blood cell count | 28 Days
Reticulocyte count | 28 days
IGF-1 | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Targeted Medical Pharma, Los Angeles, California, United States